CLINICAL TRIAL: NCT04452370
Title: Oral Etoposide Combined With Anlotinib in Advanced Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2225
Record Dates: First submitted 2020-06-11; First posted 2020-06-30 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Etoposide; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oral Etoposide+Anlotinib (Experimental): anlotinib 12mg qd, d1-14，21days/cycle oral etoposide 75mg qd，d1-10，21days/cycle
  Interventions: Drug: oral etoposide + anlotinib

INTERVENTIONS:
Drug: oral etoposide + anlotinib — anlotinib 12mg qd, d1-14，21days/cycle oral etoposide 75mg qd，d1-10，21days/cycle
  Other Names: there is no other intervention name

SUMMARY:
The hypothesis of this study is to discover if the oral Etoposide plus Anlotinib can shrink or slow the growth of pretreated advanced TNBC.

It is a single-arm, multicenter phase II clinical study of oral etoposide combined with antinib in the treatment of recurrent or metastatic triple-negative breast cancer

DETAILED DESCRIPTION:
It is a single-arm, multicenter phase II clinical study of oral etoposide combined with antinib in the treatment of recurrent or metastatic triple-negative breast cancer.

The hypothesis of this study is to discover if the oral Etoposide plus Anlotinib can shrink or slow the growth of pretreated advanced TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 year-old women; TNBC
* ECOG score: 0-1, expected survival time ≥ 3months;
* Pathologically or cytologically confirmed breast cancer;
* Anthracycline- / taxane- pretreated (adjuvant, neoadjuvant) breast cancer patients who have failed from 1-3 standard chemotherapies after recurrence and metastasis;
* According to RECIST 1.1, exist at least ≥1 measurable lesion(CT >1cm，other examination >2cm);
* The patients have enough organ function. The laboratory test indexes must comply with the following requirements:

  * Blood routine: neutrophil≥1.5G/L, platelet count ≥80G/L, hemoglobin ≥90g/L
  * Liver function: serum bilirubin ≤ 1.5 times the upper limit of normal value; ALT and AST≤2.5 times the upper limit of normal value; ALT and AST≤5 times the upper limit of normal value when liver metastasis
  * Renal function: serum creatinine ≤ 1.0times the upper limit of normal value, creatinine clearance >50ml/min（Cockcroft-Gault formula)
* Women of child-bearing age should be carried out pregnancy test (serum or urine) within 7 days before recruit, the results should be negative; and are willing to adopt the appropriate methods of contraception during the trial and 8 weeks after last administration；
* Can swallow oral drugs;
* The patients have good compliance to the therapy and follow-up to be scheduled and are able to understand the study protocol and sign the Informed Consent Form.

Exclusion Criteria:

* The patients in pregnancy or lactation growth period and did not take effective contraception;
* The patients who received ≥4 chemotherapies after recurrence and metastasis; involved in other clinical trials four weeks prior to the start of the study;
* The patients with a variety of factors that affect the oral administration and absorption of drugs;
* Prior treatment with etoposide or antiangiogenic TKI (subjects with prior use of antiangiogenic macromolecules such as bevacizumab are allowed to be enrolled);
* The patients have uncontrollable mental illness；
* Serous cavity effusion (such as pleural effusion and ascites) with clinical symptoms requiring clinical intervention or stable time less than 4 weeks;
* The patients who had serious adverse effect to oral etoposide or were allergic to etoposide.
* The patients who have only bone metastasis without other measurable lesion;
* The patients experience severe cardiovascular diseases;
* The patients experience severe upper gastrointestinal ulcer or malabsorption syndrome.
* Abnormal bone marrow functions(neutrophil<1.5G/L, platelet count <75G/L, hemoglobin <90g/L);
* Abnormal renal function(serum creatinine > 1.5 times the upper limit of normal value);
* Abnormal liver function(serum bilirubin ≤ 1.5 times the upper limit of normal value);
* The patients have uncontrollable brain metastasis;
* Active or uncontrolled infection requiring systematic treatment (except simple urinary tract infection or upper respiratory tract infection) during the 2 weeks or 2 weeks prior to enrollment;
* Previous or concurrent history of other malignant tumors.Except for the cured skin basal cell carcinoma and cervical carcinoma in situ;
* The patients do have good compliance to the therapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-07-11 (Estimated); Study Completion 2023-07-11 (Estimated)

PRIMARY OUTCOMES:
objective response rate（ORR） | up to 1 year after the last patient enrolled
  The ORR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Progression free survival（PFS） | up to 1 year after the last patient enrolled
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause
Incidence and Severity of adverse events | approximately 1.5 years
  hematologic，hepatotoxicity，Incidence of hypertension，Incidence of proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital. Chinese Academy of Medical Sciences, Beijing, China